CLINICAL TRIAL: NCT04643405
Title: An Open Label, Multiple Centers Phase Ib/II Study of APG-1387 Plus Chemotherapy in Advanced Pancreatic Adenocarcinoma
Brief Title: APG-1387 Plus Chemotherapy in Advanced Pancreatic Adenocarcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company Strategy
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APG1387PC101
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Advanced Pancreatic Cancer
Keywords: IAP inhibitor; APG-1387; Pancreatic cancer; Inhibitor of apoptosis
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — APG-1387; Injections; Gemcitabine; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- APG1387 in combination with Gemcitabine and Nab-Paclitaxel (Experimental)
  Interventions: Drug: APG-1387 for Injection; Drug: Gemcitabine; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: APG-1387 for Injection — APG1387 will be administered IV days 1， 8, 15 and 22 of a 28 day cycle.
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 will be administered IV days 1, 8, and 15 of a 28 day cycle.
Drug: Nab paclitaxel — Nab-Paclitaxel 125mg/m^2 will be administered IV days 1, 8, and 15 of a 28 day cycle.

SUMMARY:
This study is a two stage study consisting of a dose escalation phase Ib and a phase II study which include subjects with previously-treated, advanced pancreatic adenocarcinoma. Dose Limiting Toxicities (DLTs) and maximum tolerated dose (MTD) of APG1387 in combination with nab-paclitaxel and gemcitabine will be evaluated in the dose escalation phase Ib. Safety and efficacy of APG1387 plus gemcitabine and nab-paclitaxel will be evaluated in phase II.

DETAILED DESCRIPTION:
The ability of tumor cells to evade apoptosis is currently a major problem in anti-tumor therapy. IAPs are an important class of apoptosis-regulating proteins. APG-1387, a potent bivalent SMAC mimetic, small molecule of IAP inhibitor, which could inhibit pancreatic cancer proliferation as monotherapy and in combination with chemotherapy through apoptosis pathway.

It's an open label, multiple centers phase Ib/II Study. Safety and tolerability of APG1387 combined with nab-paclitaxel and gemcitabine will be evaluated in phase Ib in previously-treated, advanced pancreatic adenocarcinoma patients. Efficacy and tolerability will be evaluated in phase II study in first line standard treatment failed metastatic pancreatic adenocarcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be ≥18 years of age at time of informed consent
2. Able to comply with the study protocol, in the investigator's judgment
3. Expected survival ≥ 3 months
4. Histology or cytology confirmed as advanced pancreatic adenocarcinoma, and:

   * Standard treatment failed or intolerant to standard treatment(Phase Ib);
   * First line standard treatment failed (Phase II).
5. ECOG 0-1;
6. Adequate organ function.
7. Subjects must have at least one measurable lesion evaluated by Computed Tomography (CT) scan on RECIST ver.1.1 at pre-treatment

Exclusion Criteria:

1. Has had chemotherapy, radiation, target or other antitumor therapy within 14 days prior to the first dose of study drug.
2. Has received an investigational agent or used an investigational device within 28 days of the first dose of study drug.
3. Has received a therapy with TNFα within 28 days of the first dose of study drug.
4. Known active central nervous system involvement.
5. Has received IAP-inhibitor before.
6. Has had major surgery within 28 days of dosing of investigational agent, or minor surgery within 14 days.
7. Patients with clinically evident Hepatitis B surface antigen (HBs) positive, Hepatitis C virus (HCV) antibody positive, Human Immunodeficiency Virus (HIV) antibody positive.
8. Pregnant or breastfeeding (lactating) women.
9. Other situations that investigator think not suit for study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) of combination therapy (Applicable for: phase Ib stage ). | 28 days.
  DLT will be graded according to NCI CTCAE Version 5.0. DLT will be defined as clinically significant drug-related adverse events during the cycle one.
Overall Response Rate (Applicable for: phase II stage) . | Up to 2 years.
  Evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 2 years.
  From date of treatment start until the date of progression or the date of death due to any cause.
Duration of Response (DOR) | Up to 2 years.
  From date of response until the date of progression.
Overall Survival (OS) | Up to 2 years.
  From date of treatment start until the date of death due to any cause.
Maximum plasma concentration (Cmax) | 28 days.
  Cmax of APG-1387 and Nab-Paclitaxel will be assessed in the patients in this study.
Area under the plasma concentration versus time curve (AUC) | 28 days.
  AUC of APG-1387 and Nab-Paclitaxel will be assessed in the patients in this study.
Adverse events | Up to 2 years.
  Adverse events (AE) and serious adverse events (SAE) will be graded according to NCI CTCAE Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, MD, PhD, Study Chair — Jiangsu Ascentage Pharma Co., Ltd.
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Shi S, Zhang J, Liu R, Gao S, Xu J, Wang W, Wei M, Li J, Liu C, Xu X, Pan W, Tian X, Men L, Wang H, Liang Z, Zhu M, Yang D, Zhai Y, Yu X. A phase 1 trial of APG-1387, an IAP antagonist, with nab-paclitaxel and gemcitabine in patients with refractory metastatic pancreatic cancer. Cell Rep Med. 2025 Oct 21;6(10):102364. doi: 10.1016/j.xcrm.2025.102364. Epub 2025 Sep 19. PMID 40975066